CLINICAL TRIAL: NCT01876719
Title: A Randomized, Double-Blind, Placebo-Controlled, Forced Titration, Proof-of-Concept Study of AR08 in the Treatment of Attention Deficit Hyperactivity Disorder in Children (Ages 6 - 17)
Brief Title: AR08 for Treatment of ADHD in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR08.001
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: ADHD
Keywords: ADHD; AR08; adrenergic receptor agonists; randomized, placebo-controlled clinical trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5 mg AR08 (Experimental): 0.5 mg AR08, QD for 7 weeks
  Interventions: Drug: AR08
- 1.0 mg AR08 (Experimental): 1.0 mg AR08, QD for 7 weeks
  Interventions: Drug: AR08
- 2.0 mg AR08 (Experimental): 2.0 mg AR08, QD for 7 weeks
  Interventions: Drug: AR08
- Placebo (Placebo Comparator): Placebo, QD for 7 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR08
  Arms: 0.5 mg AR08; 1.0 mg AR08; 2.0 mg AR08
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, multiple dose, randomized, double-blind, placebo-controlled, forced titration study. Patients will be randomized to 1 of 4 treatment groups in a 1:1:1:1 ratio. One-hundred twenty (120) patients are planned to be randomized. Each patient will receive AR08 (0.5, 1, or 2 mg per day) or matching placebo for seven (7) weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV-TR criteria for a primary diagnosis of ADHD based on structured clinical interview, MINI-KID, as assessed by the Investigator
2. Minimum score of 28 on the ADHD-RS-IV at Baseline
3. Male or female ages 6 - 17 years, inclusive, at the time of Screening
4. Weighs ≥21 kg (46 pounds).
5. Is functioning at age appropriate levels intellectually, as deemed by the Investigator.

Exclusion Criteria:

1. Has a comorbid psychiatric diagnosis (comorbid psychiatric diagnosis will be established by the MINI-KID interview).
2. Has a positive response to either question 4 or 5 of the Baseline /Screening version of the pediatric Columbia Suicide Severity Rating Scale (C-SSRS)
3. History of daily usage (at least 28 days/month) of either anti-hypertensive or prophylactic anti-migraine medications prior to Screening
4. Current usage of medications known to cause QTc prolongation or ADHD medications.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ADHD-RS-IV | Day 35
  The primary endpoint is the ADHD-RS-IV; change from Baseline to Visit 7 (Day 35).

SECONDARY OUTCOMES:
CGI-ADHD-S/I | Day 35
  CGI-ADHD-S (severity) and I (improvement) - change from Baseline.
Conners' Parent Rating Scale | Day 49
  Conners' Parent Rating Scale (CPRS-R-S) will be assessed through Day 49.
Columbia Suicide Severity Rating Scale (C-SSRS) | Day 49
  Columbia Suicide Severity Rating Scale (C-SSRS) - incident rate will be assessed through Day 49.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Downey, MD, Study Director — Arbor Pharmaceuticals
Locations (13):
- United States (13):
  - Florida Clinical Research Center, LLC, Brandenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - CNS Healthcare, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Midwest Research Group at St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - CNS Healthcare, Memphis, Tennessee
  - Bayou City Research Ltd., Houston, Texas
  - Houston Clinical Trials, Houston, Texas
  - Neuroscience Associates, Herndon, Virginia